CLINICAL TRIAL: NCT04592718
Title: The Effects of Four-week Breathing Interventions on Gastrointestinal Symptoms, Heart Rate Variability, and Psychological Measures in Runners
Brief Title: Four-week Breathing Interventions on Gut Symptoms, Heart Rate Variability, and Psychological Measures in Runners
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Old Dominion University (Other)
Responsible Party: Principal Investigator, Patrick Wilson, PhD, Associate Professor of Exercise Science, Old Dominion University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Basic Science
Other Study IDs: 1655312
Record Dates: First submitted 2020-10-12; First posted 2020-10-19 (Actual); Last update posted 2021-09-09 (Actual); Status verified 2021-09

CONDITIONS: Gastrointestinal System--Abnormalities; Anxiety; Visceral Pain
MeSH Terms: conditions — Anxiety Disorders; Visceral Pain

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Slow deep breathing plus breath counting (Experimental): Participants in this group will do a daily 5-min slow deep breathing exercise (6 breaths/minute) and will also count their breaths
  Interventions: Behavioral: Slow deep breathing plus breath counting
- Normal-paced breathing plus breath counting (Active Comparator): Participants in this group will do a daily 5-min normal-paced breathing (15 breaths/minute) and will also count their breaths
  Interventions: Behavioral: Normal-paced breathing plus breath counting
- Control (No Intervention): Participants in this group will serve as a control and will not do any breathing exercises or breath counting.

INTERVENTIONS:
Behavioral: Slow deep breathing plus breath counting — Participants will perform a daily 5-min slow deep breathing exercise for 4 weeks. A breathing rate of 6 breaths per minute will be targeted. In addition, participants will count their breaths during the exercise.
  Arms: Slow deep breathing plus breath counting
Behavioral: Normal-paced breathing plus breath counting — Participants will perform a daily 5-min normal-paced breathing exercise for 4 weeks. A breathing rate of 15 breaths per minute will be targeted. In addition, participants will count their breaths during the exercise.
  Arms: Normal-paced breathing plus breath counting

SUMMARY:
Recent research has suggested that stress and anxiety levels are associated with gastrointestinal (GI) symptoms in endurance athletes (runners, cyclists, triathletes). Yet, there has been limited attempt to evaluate whether GI symptoms during running can be mitigated by interventions designed to reduce stress and anxiety. Thus, this study will evaluate the effects of four-week slow deep breathing and mindful breath counting interventions on subjective and objective measures of stress/anxiety and GI symptoms in runners with mild-to-high anxiety and that are prone to GI symptoms during runs.

ELIGIBILITY:
Inclusion Criteria:

* At least 18 years of age
* Run at least 15 miles per week
* Access to internet
* Access to a smart phone that is compatible with iOS or Android applications
* Score at least a 5 on the GAD-7
* Report to have experienced GI symptoms "sometimes", "often" or "always" during runs in the previous month.
* If on a psychotropic medication, must be on a stable dose for the past 3 months.
* Live within the contiguous United States

Exclusion Criteria:

* Younger than 18 years
* Run less than 15 miles per week
* Do not have access to the internet
* Do not have access to a smart phone that is compatible with iOS or Android applications
* Score less than 5 on the GAD-7
* Report to have "never" or "rarely" experienced GI symptoms during runs in the previous month
* Are being prescribed a psychotropic medication and have not had a stable dose for at least three months.
* Do not live within the contiguous United States

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 63 (Actual)
Dates: Start 2020-10-20 (Actual); Primary Completion 2021-06-30 (Actual); Study Completion 2021-06-30 (Actual)

PRIMARY OUTCOMES:
Change in gastrointestinal symptom occurrence | The intervention will last 4 weeks. Gastrointestinal symptoms will be collected for a 1-week period before the intervention and during the 4th week of the intervention.
  Percentage of training runs that runners experience at least 1 gastrointestinal symptom (>2 on 0-10 scale).
Change in anxiety levels | The intervention will last 4 weeks. The General Anxiety Disorder-7 will be assessed before the intervention begins, 2 weeks into the intervention, and at the end of the intervention.
  Levels of anxiety will be assessed with the General Anxiety Disorder-7 questionnaire. Scores on the General Anxiety Disorder-7 range from 0 to 21, with higher scores indicating higher levels of anxiety.

SECONDARY OUTCOMES:
Change in visceral sensitivity | The intervention will last 4 weeks. The Visceral Sensitivity Index will be assessed before the intervention begins, 2 weeks into the intervention, and at the end of the intervention.
  Perceptions of visceral sensitivity will be assessed via the Visceral Sensitivity Index. Scores on the Visceral Sensitivity Index can range from 0 to 75, with higher scores indicating a higher level of visceral sensitivity.
Change in mindfulness | The intervention will last 4 weeks. The Five Facet Mindfulness Questionnaire will be assessed before the intervention begins, 2 weeks into the intervention, and at the end of the intervention.
  Perceptions of mindfulness will be assessed via the 15-item Five Facet Mindfulness Questionnaire. Scores on the Five Facet Mindfulness Questionnaire can range from 15-75, with higher scores indicating higher levels of mindfulness.
Change in body vigilance | The intervention will last 4 weeks. The Body Vigilance Scale will be assessed before the intervention begins, 2 weeks into the intervention, and at the end of the intervention.
  Perceptions of body vigilance will be assessed via the Body Vigilance Scale. Scores on the Body Vigilance Scale can range from 0-40, with higher levels meaning greater amounts of body vigilance.
Change in heart rate variability (Ln RMSSD) | The intervention will last 4 weeks. Ln RMSSD will be assessed before the intervention begins, and at the end of the intervention.
  Heart rate variability will be assessed via a portable fingertip monitor (CorSense) and quantified as the Ln root mean square of successive differences (Ln RMSSD) between normal heartbeats.

CONTACTS AND LOCATIONS:
Overall Officials: Patrick Wilson, Principal Investigator — Old Dominion University
Locations (1):
- Human Performance Laboratory, Norfolk, Virginia, United States

IPD SHARING:
Plan to Share IPD: No